CLINICAL TRIAL: NCT04583696
Title: The Investigation of Effect on Blood Lipid Parameters With Walnut Addition of Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Sifa University (Other)
Responsible Party: Principal Investigator, Fatih Cesur, Principal Investigator, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 227-63
Record Dates: First submitted 2020-09-22; First posted 2020-10-12 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Risk Factor
Keywords: cholesterol; walnut consumption; small dense LDL; blood lipids; dietary fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walnut Consumption of Healthy Volunteers (Experimental)
  Interventions: Dietary Supplement: The Investigation of effect on Blood Lipid parameters with walnut addition of Diet

INTERVENTIONS:
Dietary Supplement: The Investigation of effect on Blood Lipid parameters with walnut addition of Diet — Participants were asked to consume 30 g of walnuts daily for 21 days. Individuals have consumed walnuts on an empty stomach in the morning or with breakfast.

SUMMARY:
Introduction There is a strong relationship between eating habits and diseases of the cardiovascular system. It is known that walnut consumption has positive effects on cardiovascular system diseases. However, its effect on small dense LDL (sdLDL) is discussed. Therefore in this study, you participated the effects of walnut consumption on the serum lipids values, especially sdLDL values of healthy volunteers.

Methods Volunteers participating in this study were offered 30 grams of walnuts per day for 21 days. Walnuts were consumed on empty stomach or with breakfast every morning for 21 days. The blood values of subjects were measured at the beginning and the end of the study. The serum was obtained from the taken blood and blood lipid/hemoglobin parameters were measured on routine blood work. Food consumption records and surveys were taken from individuals.

ELIGIBILITY:
Inclusion Criteria:

* Do not consume any products such as nuts and walnuts (the frequency of consumption should not be more than once a week)
* Have no allergies to foods such as nuts and walnuts
* Do not take drugs on a daily and continuous basis

Exclusion Criteria:

* Obesity
* Diabetes Mellitus
* Acoholic and chronic diseases such as kidney
* Thyroid
* Hepatitis
* Cancer etc.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2015-03-10 (Actual); Study Completion 2015-04-24 (Actual)

PRIMARY OUTCOMES:
Blood from the participants was collected before and at the end of the study. Later in this study, sdLDL levels of blood taken from participants were measured by the Elisa method. | Within research completion, an average of 2 week
  It can be said that walnut consumption reduces the risk of CAD. In 30% of patients taking cholesterol-lowering drugs, cholesterol parameters may drop to the desired levels and severe vascular lesions still may occur. Also, individuals with normal LDL values may have cardiovascular diseases. Findings are suggesting that in these individuals, the prevalence of CAD is higher due to sdLDL positivity. sdLDL passes through the endothelial barrier easier and is exposed to oxidation more than LDL, which is larger and lower in density. Therefore is atherogenic.
Blood from the participants was collected before and at the end of the study. Later, the serum lipids of the blood taken from the participants consuming walnuts were measured in the hospital. | The first day of the research and the end day (3 weeks later) were analyzed.
  It can be said that walnut consumption reduces the risk of CAD. The fact that walnuts contain fatty acids can be shown as a reason for their beneficial effect on blood lipid levels. We can attribute this to the fact that walnuts contain high levels of unsaturated and low levels of saturated fatty acids. In various studies, the walnut-enriched diet has been reported to reduce TC, LDL, and TG

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iwamoto M, Imaizumi K, Sato M, Hirooka Y, Sakai K, Takeshita A, Kono M. Serum lipid profiles in Japanese women and men during consumption of walnuts. Eur J Clin Nutr. 2002 Jul;56(7):629-37. doi: 10.1038/sj.ejcn.1601400. PMID 12080402
- [Result] Jenkins DJA, Kendall CWC, Lamarche B, Banach MS, Srichaikul K, Vidgen E, Mitchell S, Parker T, Nishi S, Bashyam B, de Souza RJ, Ireland C, Pichika SC, Beyene J, Sievenpiper JL, Josse RG. Nuts as a replacement for carbohydrates in the diabetic diet: a reanalysis of a randomised controlled trial. Diabetologia. 2018 Aug;61(8):1734-1747. doi: 10.1007/s00125-018-4628-9. Epub 2018 May 23. PMID 29789878
- [Result] Ai M, Otokozawa S, Asztalos BF, Ito Y, Nakajima K, White CC, Cupples LA, Wilson PW, Schaefer EJ. Small dense LDL cholesterol and coronary heart disease: results from the Framingham Offspring Study. Clin Chem. 2010 Jun;56(6):967-76. doi: 10.1373/clinchem.2009.137489. Epub 2010 Apr 29. PMID 20431054
- [Result] Mohammadi-Sartang M, Bellissimo N, Totosy de Zepetnek JO, Bazyar H, Mahmoodi M, Mazloom Z. Effects of walnuts consumption on vascular endothelial function in humans: A systematic review and meta-analysis of randomized controlled trials. Clin Nutr ESPEN. 2018 Dec;28:52-58. doi: 10.1016/j.clnesp.2018.07.009. Epub 2018 Sep 1. PMID 30390893
- [Result] Bamberger C, Rossmeier A, Lechner K, Wu L, Waldmann E, Stark RG, Altenhofer J, Henze K, Parhofer KG. A Walnut-Enriched Diet Reduces Lipids in Healthy Caucasian Subjects, Independent of Recommended Macronutrient Replacement and Time Point of Consumption: a Prospective, Randomized, Controlled Trial. Nutrients. 2017 Oct 6;9(10):1097. doi: 10.3390/nu9101097. PMID 28984822